CLINICAL TRIAL: NCT00805792
Title: Mayo Acute Stroke Trial for Enhancing Recovery
Acronym: MASTER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, James F. Meschia, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-005098
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Results first posted 2012-11-14 (Estimated); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke; treatment; recovery; donepezil; Aricept
MeSH Terms: conditions — Ischemic Stroke | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Donepezil (Experimental): Participants received treatment with donepezil within 24 hours after the onset of ischemic stroke symptoms. Participants received donepezil 5 mg/day for 30 days, followed by an increase to 10 mg/day for 60 days.
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — Study participants will be treated with donepezil orally at an initial dose of 5 mg daily for the first 4 weeks, then increased at their 30-day visit by 5 mg to a maximum dose of 10 mg daily, if tolerated. If the participant does not tolerate the 10 mg dose, they will remain on 5 mg through the course of the study.
  Other Names: Aricept

SUMMARY:
This study involves treating patients that have suffered an acute ischemic stroke with the medication donepezil (Aricept ®). The hypothesis is that taking donepezil (FDA-approved for the treatment of Alzheimer's Disease) for the first 90 days following a stroke enhances recovery.

DETAILED DESCRIPTION:
We hypothesize that donepezil (5 mg per day, titrated up to 10 mg per day as tolerated) will enhance recovery following stroke by improving attention, learning and memory thereby enhancing rehabilitation. The null hypothesis is that the probability of a favorable outcome among post-stroke donepezil users is equal to that observed among similar participants in an existing National Institutes of Neurological Disorders and Stroke (NINDS) resource, the Phase III clinical trial of Tissue Plasminogen Activator (tPA) for acute ischemic stroke. The NINDS tPA stroke trial has been used as historical control data in pilot trials of reperfusion and neuroprotection.

The MASTER trial will be a multicenter, single-arm NINDS Recominant tPA trial-controlled, modified 2-stage adaptive clinical trial set in 2 tertiary care hospitals in the United States. Participants will be men and women with acute (< 24 hours of onset of symptoms) ischemic stroke. A favorable outcome will be defined as National Institutes of Health Stroke Scale (NIHSS) values of 0 or 1 at 90 days post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* Definite or probable acute ischemic cerebrovascular syndrome (AICS), as defined by Kidwell et al (Stroke. 2003;34:2995-8).
* Experimental treatment started within 24 hours of onset of symptoms.
* Age ≥ 18 years.
* Ability and willingness to return for follow-up visits.
* Willingness of an available informant who knows the patient well to participate in informant-based questionnaires for the duration of the follow-up period.
* Living in independent or semi-independent living situation before the stroke.
* Fluent in English before the stroke.
* Provides written informed consent.
* Near visual acuity of at least 20/200 in at least one eye.
* Auditory acuity of at least having the ability to detect finger rubbing in at least one ear.

Exclusion Criteria:

* Parkinson's disease or restless leg syndrome.
* Partial or generalized seizures.
* No acute decompensated heart failure
* Routinely requiring daytime supplemental oxygen before the stroke; study participants on continuous positive air pressure (CPAP) for obstructive sleep apnea remain eligible.
* Gastrointestinal or genitourinary surgery within 1 month of screening.
* Gastrointestinal bleeding.
* Syncope or symptomatic bradycardia.
* Creatinine ≥ 3.5 mg/dL or requiring dialysis.
* Peptic ulcer disease.
* Asthma.
* Tracheostomy or endotracheal intubation.
* Taking donepezil or other acetylcholinesterase inhibitor at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F. Meschia, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Background] Meschia JF, McNeil RB, Barrett KM, Brott TG, Graff-Radford NR, Brown RD Jr. Mayo Acute Stroke Trial for Enhancing Recovery (MASTER) protocol. J Stroke Cerebrovasc Dis. 2010 Jul-Aug;19(4):299-310. doi: 10.1016/j.jstrokecerebrovasdis.2009.05.005. PMID 20610186
- [Background] National Institute of Neurological Disorders and Stroke rt-PA Stroke Study Group. Tissue plasminogen activator for acute ischemic stroke. N Engl J Med. 1995 Dec 14;333(24):1581-7. doi: 10.1056/NEJM199512143332401. PMID 7477192
- [Result] Barrett KM, Brott TG, Brown RD Jr, Carter RE, Geske JR, Graff-Radford NR, McNeil RB, Meschia JF; Mayo Acute Stroke Trial for Enhancing Recovery (MASTER) Study Group. Enhancing recovery after acute ischemic stroke with donepezil as an adjuvant therapy to standard medical care: results of a phase IIA clinical trial. J Stroke Cerebrovasc Dis. 2011 May-Jun;20(3):177-82. doi: 10.1016/j.jstrokecerebrovasdis.2010.12.009. Epub 2011 Feb 3. PMID 21295494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment extended from November 2008 through April 2010. The study was conducted at the Mayo Clinic sites in Jacksonville, FL and Rochester, MN.
Period: Overall Study
Arm/Group | Donepezil
Started | 33
Completed | 28
Not Completed | 5
Not completed — Death | 3
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Donepezil
Number analyzed (Participants) | 33
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [54 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 33
Number of Participants with Previous Ischemic Stroke [Number; unit: participants]
  Previous ischemic stroke | 5
  No previous ischemic stroke | 28
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 27.1 [24.7 to 30.6]
Participant Scores on National Institutes of Health Stroke Scale [Number; unit: participants] — The National Institutes of Health Stroke Scale (NIHSS) is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The range of scores is from 0 (normal) to 42 (profound effect of stroke on patient).
  participants
    Mild (<6) | 16
    Moderate (6-13) | 12
    Severe (>13) | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With National Institutes of Health Stroke Scale (NIHSS) Score = 0 or 1 at Day 90
Description: The National Institutes of Health Stroke Scale (NIHSS) is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The range of scores is from 0 (normal) to 42 (profound effect of stroke on patient).
Time Frame: 90 days post-stroke
Population: Intention-to-treat analysis, all treated participants (n=33). Unobserved because of death (n=3) or loss to follow up (N=2) treated as nonresponse.
Measure: Number; unit: percentage of participants
Arm/Group | Donepezil
Number analyzed (Participants) | 33
percentage of participants
  Stroke severity (NIHSS) mild (<6) (n=11/16) | 69
  Stroke severity (NIHSS) moderate (6-13) (n=4/12) | 33
  Stroke severity (NIHSS) severe (>13) (n=0/5) | 0
  Overall (n=15/33) | 45

2. Secondary Outcome: Change in Mean National Institutes of Health Stroke Scale (NIHSS) Score at 90 Days Post-stroke
Description: as for outcome 1
Time Frame: baseline, 90 days post-stroke
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Donepezil
Number analyzed (Participants) | 33
units on a scale | -2.8 (0.8)
Statistical Analysis 1: Comparison: Donepezil; The statistical significance of the change was assessed by the P value associated with estimated regression coefficient (beta coefficient or slope); Test type: Superiority or Other; p < .001, Regression, Linear

3. Secondary Outcome: Change in Mean Barthel Index of Activities of Daily Living Score at 90 Days Post-stroke
Description: The Barthel Index of Activities of Daily Living (ADLs) measures functional disability by quantifying patient performance in 10 activities of daily life. These activities can be grouped according to self-care (feeding, grooming, bathing, dressing, bowel and bladder care, and toilet use) and mobility (ambulation, transfers, and stair climbing). 5-point increments are used in scoring, with a maximal score of 100 indicating that a patient is fully independent in physical functioning, and a lowest score of 0 representing a totally dependent bed-ridden state.
Time Frame: baseline, 90 days post-stroke
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Donepezil
Number analyzed (Participants) | 33
units on a scale | 21.4 (5.2)
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .001, Regression, Linear

4. Secondary Outcome: Change in Mean Score on Mini Mental State Exam at 90 Days Post-stroke
Description: The mini-mental state examination (MMSE) is a 30-point questionnaire test that is used to screen for cognitive impairment. The questionnaire samples functions including arithmetic, memory and orientation to time and place. Scores range from 0 to 30. Any score greater than or equal to 25 points is effectively normal (intact). Below this, scores can indicate severe (≤9 points), moderate (10-20 points) or mild (21-24 points) cognitive impairment.
Time Frame: baseline, 90 days post-stroke
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Donepezil
Number analyzed (Participants) | 33
units on a scale | 4.4 (1.2)
Statistical Analysis 1: Comparison: Donepezil; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .001, Regression, Linear

5. Secondary Outcome: Change in Time to Complete Neuropsychological Trail Making Tests A and B at 90 Days Post-stroke
Description: The Trail-making test consists of two parts in which the subject is instructed to connect a set of 25 dots as fast as possible while still maintaining accuracy. It can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning. There are two parts to the test: A, in which the targets are all numbers (1,2,3, etc.)and the test taker needs to connect them in sequential order, and B, in which the subject alternates between numbers and letters (1, A, 2, B, etc.).
Time Frame: baseline, 90 days post-stroke
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Donepezil
Number analyzed (Participants) | 33
seconds
  Trail Making Test A | -43.4 (9.2)
  Trail Making Test B | -67.3 (13.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 90-day course of therapy.
Arm/Group | Donepezil
Serious Adverse Events (participants affected / at risk) | 10/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=33)
Death (General disorders) | 3 (3)
Recurrent stroke (Vascular disorders) | 2 (2)
Transient ischemic attack (Vascular disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Carotid angioplasty and stent placement (Vascular disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Chest pain/leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=33)
Fatigue (General disorders) | 17 (17)
Insomnia (General disorders) | 16 (16)
Depression (Psychiatric disorders) | 13 (13)
Nausea (Gastrointestinal disorders) | 11 (11)
Loss of appetite (Gastrointestinal disorders) | 10 (10)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes